CLINICAL TRIAL: NCT01276106
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Phase II Study of AC-201 in Patients With Type 2 Diabetes Mellitus
Brief Title: Study of AC-201 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-201-DM-001
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: AC-201; Interleukin 1 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — diacerein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC-201, 25mg (Experimental): 25mg BID for 24 weeks
  Interventions: Drug: AC-201, 25mg
- AC-201, 50mg (Experimental): 50mg BID for 24 weeks
  Interventions: Drug: AC-201, 50mg
- AC-201, 75mg (Experimental): 75mg BID for 24 weeks
  Interventions: Drug: AC-201, 75mg
- Placebo (Placebo Comparator): Placebo BID for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-201, 25mg — Capsule, 25mg BID
  Arms: AC-201, 25mg
Drug: AC-201, 50mg — Capsule, 50mg BID
  Arms: AC-201, 50mg
Drug: AC-201, 75mg — Capsule, 75mg BID
  Arms: AC-201, 75mg
Drug: Placebo — Placebo BID
  Arms: Placebo

SUMMARY:
This is a 24-week randomized placebo-controlled study to investigate the effect of an oral IL-1beta inhibitor AC-201 in patients with type 2 diabetes mellitus already treated on different background diabetes therapies.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of the study procedures and agreement to participate in the study by giving written informed consent
* Males and females age 20 to 75 years, inclusive
* HbA1c ≥7.5% and ≤10%
* BMI ≤45 kg/m2
* FPG ≤270 mg/dL
* Diagnosis of type 2 diabetes mellitus for ≥6 months
* On a stable regimen of oral anti-diabetic medications for ≥3 months
* Willingness to maintain stable diet and exercise throughout the study
* Willingness to maintain current doses/regimens of vitamins and dietary supplements throughout the study
* Female patients of childbearing potential and female partners of male patients must be willing to use adequate contraception during the study. All females of childbearing potential must have a negative urine pregnancy test at screening.

Exclusion Criteria:

* History of type 1 diabetes and/or history of ketoacidosis
* History of diabetic neuropathy resulting in significant functional impairment and/or requiring active medical or surgical management, including chronic pain syndromes, gastroparesis, skin ulceration, or amputation
* History of long-term therapy with insulin (>30 days) within 1 year of screening;
* Pregnancy or lactation
* Current treatment with any of the following medications within 2 months of screening
* Anti inflammatory drugs, including chronic daily use of systemic corticosteroids (aspirin ≤325 mg per day is allowed)
* IL-1 modulators: anakinra and rilonacept
* Immunosuppressive drugs: TNF inhibitors and IL-6 monoclonal antibody
* History of severe hypoglycemic episodes within 6 months of screening
* Hypersensitivity to AC-201 or anthraquinone derivatives
* Surgery within 30 days prior to screening
* Serum creatinine >1.5 mg/dL for males or >1.4 mg/dL for females
* Presence of cancer or history of cancer within the past 5 years other than basal or squamous cell carcinoma of the skin and carcinoma in situ of the cervix
* Advanced stage heart failure: New York Heart Association Class III or IV cardiac status or hospitalization for congestive heart failure
* History of unstable angina, myocardial infarction, uncontrolled arrhythmias, cerebrovascular accident, transient ischemic attack, or any revascularization, including percutaneous transluminal coronary angioplasty, within 6 months of screening
* Uncontrolled hypertension (defined as systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg on ≥3 assessments at screening)
* Known to be infected with human immunodeficiency virus (HIV)
* History of acquired immune deficiency syndrome
* History of TB, active TB (pulmonary, extra-pulmonary, or military), or a positive test for TB confirmed by a PA chest x-ray within 6 months prior to screening
* History of acute infection with Epstein-Barr Virus (EBV), cytomegalovirus (CMV), or hepatitis C virus (HCV) within 4 weeks prior to screening
* History of chronic active (not latent) hepatitis B virus, HCV, or CMV infection;
* History of drug or alcohol abuse
* Aspartate aminotransferase >3 × the upper limit of normal (ULN) or alanine aminotransferase >3 × ULN at screening
* Total bilirubin >1.5 × ULN at screening
* Triglycerides >500 mg/dL at screening
* Poor mental function or any other reason to expect patient difficulty in complying with the study requirements
* Acute infections that may affect blood glucose control within 4 weeks prior to screening
* Known bilateral renal artery stenosis, patient with a solitary kidney, or a post renal transplant
* History of autoimmune disease or collagen vascular disease
* History of hyperthyroidism or hypocorticism
* Participation in any AC-201 studies within 1 year prior to screening
* Participation in an investigational drug study within 30 days prior to screening
* Any other serious diseases which, in the opinion of the investigator, might pose a risk to the patient or make participation not in the patient's best interest.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - Catalina Research Institute, LLC, Chino, California
  - National Research Institute, Los Angeles, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Midwest Institute for Clinical Research, Inc., Indianapolis, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - PriMed Clinical Research, Kettering, Ohio
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Cheng Ching General Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Kuang Tien General Hospital, Taichung
  - Cardinal Tien Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Tri-Service General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited in 21 study centers, which were located in 2 countries (USA and Taiwan)
Groups:
- AC-201, 25mg BID: AC-201: Capsule, 25mg BID
- AC-201, 50mg BID: AC-201: Capsule, 50mg BID
- AC-201, 75mg BID: AC-201: Capsule, 75mg BID
- Placebo: Placebo: Capsule, BID
Period: Overall Study
Arm/Group | AC-201, 25mg BID | AC-201, 50mg BID | AC-201, 75mg BID | Placebo
Started | 65 | 64 | 65 | 65
Completed | 53 | 55 | 49 | 52
Not Completed | 12 | 9 | 16 | 13
Not completed — Adverse Event | 3 | 3 | 11 | 3
Not completed — Withdrawal by Subject | 6 | 3 | 1 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 2
Not completed — Insufficient therapeutic effects | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline was defined as the last measurement obtained on or before the first dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-201, 25mg BID | AC-201, 50mg BID | AC-201, 75mg BID | Placebo | Total
Number analyzed (Participants) | 65 | 64 | 65 | 65 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 55 (9) | 57 (9) | 55 (8) | 56 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 27 | 33 | 131
  Male | 27 | 31 | 38 | 32 | 128
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 38 | 37 | 150
  Taiwan | 27 | 27 | 27 | 28 | 109
HbA1c [Mean (Standard Deviation); unit: %] | 8.4 (0.6) | 8.3 (0.7) | 8.5 (0.7) | 8.4 (0.7) | 8.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Description: For efficacy analyses, the primary analysis was at Week 24 Endpoint, defined as the last valid post-baseline measurement taken at or before Week 24. Efficacy results for treatment groups were considered statistically significant if change from baseline relative to placebo had p<0.05.
Time Frame: 24 weeks
Population: The Full Analysis Set included all randomized patients who received at least 1 dose of study drug and had a baseline and at least 1 post-baseline HbA1c assessment.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | AC-201, 25mg BID | AC-201, 50mg BID | AC-201, 75mg BID | Placebo
Number analyzed (Participants) | 63 | 61 | 62 | 63
percentage points | 0.03 (0.123) | -0.07 (0.126) | -0.13 (0.125) | 0.22 (0.123)
Statistical Analysis 1: Comparison: AC-201, 75mg BID vs Placebo; Change from baseline in HbA1c was analyzed using an analysis of covariance model with change in HbA1c as the dependent variable, treatment as a fixed effect, and baseline HbA1c as a covariate; Test type: Superiority or Other; p = 0.044, ANCOVA — No adjustments for multiple comparisons were made and a value of p<0.05 was considered statistically significant; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.70 to -0.01], Standard Error of Mean 0.175
Statistical Analysis 2: Comparison: AC-201, 50mg BID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0979, ANCOVA — No adjustments for multiple comparisons were made and a value of p<0.05 was considered statistically significant; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.64 to 0.05], Standard Error of Mean 0.176
Statistical Analysis 3: Comparison: AC-201, 25mg BID vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2643, ANCOVA — No adjustments for multiple comparisons were made and a value of p<0.05 was considered statistically significant; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.54 to 0.15], Standard Error of Mean 0.174

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | AC-201, 25mg BID | AC-201, 50mg BID | AC-201, 75mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 3/65 | 2/64 | 2/65 | 1/65
Other Adverse Events (participants affected / at risk) | 19/65 | 25/64 | 38/65 | 15/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-201, 25mg BID (N=65) | AC-201, 50mg BID (N=64) | AC-201, 75mg BID (N=65) | Placebo (N=65)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Ulcer Hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Breast Cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Urinary Incontenence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AC-201, 25mg BID (N=65) | AC-201, 50mg BID (N=64) | AC-201, 75mg BID (N=65) | Placebo (N=65)
Diarrhea (Gastrointestinal disorders) | 12 (14) | 10 (12) | 21 (25) | 6 (7)
Upper respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 10 (14) | 4 (4) | 6 (6)
Chromatouria (Renal and urinary disorders) | 2 (2) | 5 (5) | 13 (13) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 2 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Back Pain (Nervous system disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less